CLINICAL TRIAL: NCT00973505
Title: Significance of CYP19 Genetic Polymorphism on Musculoskeletal Symptom & Complication of Aromatase Inhibitor(AI)
Brief Title: CYP19 Genetic Polymorphism & Aromatase Inhibitor(AI)
Acronym: AI-CYP19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Korea University (Other)
Responsible Party: Eun Sook, Lee, Korea University Anam Hospital
Other Study IDs: AN09021
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Breast Neoplasms; Arthralgia; Arthritis; Genetic Polymorphism
Keywords: Breast neoplasms; Aromatase inhibitors; Genetic polymorphisms; Arthralgia; Arthritis
MeSH Terms: conditions — Breast Neoplasms; Arthralgia; Arthritis | interventions — Anastrozole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CYP19: CYP19 genetic polymorphism
  Interventions: Drug: Aromatase Inhibitor(Femara or Arimidex)

INTERVENTIONS:
Drug: Aromatase Inhibitor(Femara or Arimidex) — Femara(Letrozole) 2.5mg 1tab qd, Arimidex(Anastrozole) 1mg 1tab qd

SUMMARY:
The purpose of this study is to investigate the relationship between the side effects(especially arthralgia and arthritis) which appear in the patients who are prescribed aromatase inhibitor(AI) and the CYP19 genetic polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must sign the informed consent.
2. The patient must sign the informed consent of genetic screening test.
3. The patient must be between 18 years old and 80 years old who can make a decision independently.
4. The patient must be post-menopause status.
5. The patient should be the stage 1,2 or 3 of the breast cancer.
6. The test result of the estrogen receptor or progesterone receptor is positive, so the patient should be taking the medication of AI (Aromatase Inhibitor).

Exclusion Criteria:

1. The patient is pre-menopause status.
2. The test result of serum FSH level is below 30mU/ml.
3. The test result of the hormone receptor(ER & PR) is negative or unknown.
4. Patient's breast cancer stage is 4 which has systemic metastatics.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients taking the medication of AI (aromatase inhibitor) in post menopause status.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Change of SNPs (PCR & sequencing), Estrogen, Inflammatory Cytokine level | 6, 12 months

SECONDARY OUTCOMES:
EORTC (European Organization for Research and Treatment of Cancer)- QOL(Quality of Life)- C30, BR23 & Skeletal pain information, BMI | 3,6,12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eun Sook Lee, MD, PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hopital, Seoul, South Korea